CLINICAL TRIAL: NCT02051075
Title: A Randomized Controlled Trial to Compare Fertilizations With Immotile Sperm After Pentoxyphylline Activation Alone, or With Chemical Oocyte Activation
Brief Title: Fertilizations With Immotile Sperm: Pentoxyphylline Activation Alone, or With Chemical Oocyte Activation
Acronym: PXN
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: failure to recruit
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Shahar Kol MD, Durector, IVF Unit, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMB 0443-13; 0443-13-RMB (Other: Rambam Medical Center)
Record Dates: First submitted 2014-01-29; First posted 2014-01-31 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Infertility
Keywords: IVF; ICSI; Asthenospermia; pentoxyphylline; Spermatozoa
MeSH Terms: conditions — Infertility; Asthenozoospermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PXN only (Active Comparator): Sperm activation with PXN before ICSI
  Interventions: Biological: PXN sperm treatment
- PXN activation and oocyte activation (Experimental): Sperm activation with PXN and oocyte activation
  Interventions: Biological: Sperm activation with PXN and oocyte activation

INTERVENTIONS:
Biological: PXN sperm treatment — immotile sperm activation with PXN
  Arms: PXN only
Biological: Sperm activation with PXN and oocyte activation
  Arms: PXN activation and oocyte activation

SUMMARY:
Immotile sperm is a rather frequent problem encountered in IVF patients. Treatment is usually based on inducing motility with pentoxyphylline (PXN) followed by ICSI. However, fertilization rate with this method is still lower compared with ICSI using motile sperm. One of the reasons for that is the immotile sperm inability to activate the oocyte Our research hypothesis is that better fertilization rate can be accomplished in these cases by combining PXN sperm activation with Ca ionophore oocyte activation.

ELIGIBILITY:
Inclusion Criteria:

* Women up to 35 years of age
* immotile sperm
* At least 6 mature eggs

Exclusion Criteria:

* globozoospermia
* "Freeze all" cycles because of OHSS risk.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy | One month post oocyte retrieval
  Demonstration of fetal heart activity 1 month post oocyte retrieval.

SECONDARY OUTCOMES:
Fertilization rate | One day post oocyte retrieval
  Normal, 2 pronuclei, zygote one day post ICSI

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam medical Center, Haifa, Israel, Israel